CLINICAL TRIAL: NCT07400900
Title: Effectiveness of a Standardised Stabilisation Exercise Protocol in Volleyball Players With Non-traumatic Shoulder Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Alberto Roldán, PhD, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VolleyShoulder
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Shoulder Instability
Keywords: voleyball; shoulder pain; instability; exercise; Derby Shoulder Instability Rehabilitation Programme; randomized controlled trial; overhead
MeSH Terms: conditions — Shoulder Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study uses an interventional, parallel-group randomized controlled design to compare a standardized shoulder stabilization exercise program with a no-treatment control condition in amateur volleyball players with atraumatic shoulder instability. Participants are randomly assigned in a 1:1 ratio to one of the two study arms. The interventional group follows a structured rehabilitation protocol based on the Derby Shoulder Instability Rehabilitation Programme, conducted three times per week for eight weeks, while the control group receives no active intervention ("wait-and-see").
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Wait and see during 8 weeks
- Intervention group (Experimental): Participants assigned to the intervention group will complete the Derby Shoulder Instability Rehabilitation Programme (DSIRP), a structured and progressive exercise-based protocol specifically designed for individuals with atraumatic shoulder instability. Participants in this arm will perform the program three times per week, 25 minutes per session, over a total of 8 weeks. The intervention is supervised by trained physiotherapists, although progression criteria remain standardized to ensure reproducibility. No adjunct treatments (manual therapy, modalities, taping, etc.) are permitted during the intervention period. This arm aims to improve pain, functional capacity, proprioceptive control, shoulder mobility, and strength in young volleyball players with atraumatic instability, following the dosage and progression described in Bateman et al. (2015) and aligned with the intervention structure detailed in the study protocol
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants assigned to the intervention group will complete the Derby Shoulder Instability Rehabilitation Programme (DSIRP), a structured and progressive exercise-based protocol specifically designed for individuals with atraumatic shoulder instability. The program integrates strengthening exercises, proprioceptive and neuromuscular control training, plyometric drills, and speed-oriented stabilization tasks. Progression through the exercises is criterion-based, following predefined functional milestones to ensure appropriate challenge and individualized adaptation.
  The DSIRP focuses on enhancing dynamic glenohumeral stability through rotator-cuff activation, scapular control, and kinetic-chain coordination. Each session includes components targeting isometric and isotonic strengthening, closed-chain stability tasks, rhythmic stabilization, rapid-response perturbation activities, and overhead-sport-specific movement patterns relevant to volleyball athletes.
  Other Names: Derby Shoulder Instability Programme
  Arms: Intervention group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of a standardized shoulder stabilization exercise program in amateur volleyball players diagnosed with atraumatic shoulder instability. Shoulder pain is one of the most prevalent musculoskeletal complaints, affecting up to two-thirds of the general population at some point in life and frequently leading to long-term symptoms, functional limitations, sleep disturbances, and high socio-economic costs. Atraumatic glenohumeral instability is particularly common among athletes performing overhead movements, such as volleyball players, who are repeatedly exposed to high-velocity external and internal rotation actions during serves and spikes.

The Derby Shoulder Instability Rehabilitation Programme (DSIRP) is a structured, reproducible protocol integrating strengthening, proprioceptive, neuromuscular control, plyometric, and speed-oriented exercises. Although widely used in clinical practice, evidence supporting its superiority over the natural progression of the condition remains limited. More than 80% of physiotherapists in the United Kingdom do not use specific standardized protocols for atraumatic shoulder instability, highlighting the need for high-quality clinical trials that evaluate structured rehabilitation approaches.

This study will recruit amateur volleyball players aged 20 to 30 years with a clinical diagnosis of atraumatic shoulder instability lasting more than 3 months. Participants will be randomized (1:1) into two parallel groups: an experimental group performing the DSIRP for 8 weeks (three 25-minute sessions per week), and a control group following a "wait-and-see" approach. Outcome measures will be assessed at baseline, 1 month, and 2 months (post-intervention). The primary outcomes include pain intensity measured with the Numeric Pain Rating Scale and shoulder disability measured with the Spanish version of the Shoulder Pain and Disability Index. Secondary outcomes include external rotation strength, grip strength, shoulder range of motion, and health-related quality of life assessed with the SF-12 questionnaire. All measurements use validated instruments with high reliability for clinical and research settings.

Statistical analysis will follow an intention-to-treat approach using mixed-model repeated-measures ANOVA or non-parametric alternatives when appropriate. Effect sizes and Bonferroni correction for multiple comparisons will be applied. An independent biostatistician blinded to allocation will conduct the analysis. The study follows CONSORT and TIDieR guidelines for reporting and intervention description.

This trial seeks to determine whether a structured, progressive stabilization protocol offers clinically meaningful improvements in pain, disability, strength, mobility, and quality of life compared with no intervention in young volleyball players with atraumatic shoulder instability. Results may support the implementation of standardized rehabilitation strategies in physiotherapy practice for this condition.

DETAILED DESCRIPTION:
Atraumatic shoulder instability is a prevalent condition among athletes who perform repetitive overhead movements, particularly volleyball players. The biomechanical demands of serving, spiking, and blocking expose the glenohumeral joint to repeated high-velocity rotational forces, which may contribute to impaired neuromuscular control, altered proprioception, and insufficient dynamic stabilization. These factors can lead to recurrent symptoms of pain, weakness, and functional limitation, often persisting for extended periods and interfering with sports performance and daily activities.

Although physiotherapy is widely recognized as a first-line approach for managing atraumatic shoulder instability, clinical practice frequently lacks standardized and reproducible rehabilitation protocols. Existing programs vary significantly in content, dosage, and progression criteria, limiting consistency across clinicians and settings. The Derby Shoulder Instability Rehabilitation Programme (DSIRP) is one of the few structured intervention models specifically designed for this condition. It integrates strengthening, proprioception, plyometric exercises, and motor control tasks, with progression based on clearly defined functional milestones. However, despite its clinical use, robust comparative evidence supporting its effectiveness remains limited.

This randomized controlled trial aims to evaluate the clinical impact of an eight-week DSIRP-based intervention compared with no active treatment in amateur volleyball players aged 20 to 30 years with at least three months of atraumatic shoulder instability. The study follows CONSORT and TIDieR recommendations to ensure transparent reporting and comprehensive intervention description. Participants are randomly allocated in a 1:1 ratio to either the experimental group, which performs the structured exercise program three times per week, or the control group, which receives no intervention ("wait-and-see"). The analytical team remains blinded to group assignment.

The intervention is designed to address multiple dimensions of shoulder stability, including rotator-cuff strength, scapular control, reactive stability, and proprioceptive acuity. It progresses through phases that incorporate isometric and isotonic strengthening, closed-chain stability tasks, rhythmic stabilization, plyometric drills, and functional movement patterns relevant to overhead athletes. Session duration and frequency are standardized, but progression criteria ensure individualized advancement according to each participant's ability to meet predefined performance targets.

Outcome assessments are conducted at baseline, one month, and after the completion of the eight-week intervention. Measures span several domains relevant to shoulder instability, including pain intensity, self-reported disability, shoulder mobility, isometric strength, and overall health-related quality of life. All clinical instruments used in the study have demonstrated strong reliability and validity in previous research. The measurement protocol ensures standardized positioning and examiner consistency to reduce variability.

The statistical analysis incorporates repeated-measures models to evaluate changes over time and between groups. Parametric or non-parametric methods are selected based on data distribution, and effect sizes are calculated to quantify the magnitude of observed changes. A blinded biostatistician performs all analyses to minimize bias.

This study is designed to generate high-quality evidence on the usefulness of a structured, pathology-specific rehabilitation program for atraumatic shoulder instability in young overhead athletes. By comparing the DSIRP-based intervention with a no-treatment control condition, the trial aims to clarify whether a well-defined and reproducible exercise protocol leads to meaningful improvements in pain, function, strength, and mobility. Findings may inform clinical practice, support the adoption of standardized rehabilitation pathways, and contribute to reducing the variability that currently characterizes conservative management of this condition.

ELIGIBILITY:
Inclusion criteria:

Amateur volleyball players. Age range: 18 to 30 years. Clinical diagnosis of atraumatic shoulder instability. Symptom duration greater than 3 months.

Exclusion criteria:

Previous surgeries on the affected shoulder. Previous fractures of the affected shoulder. History of traumatic shoulder dislocation. Shoulder pain originating from cervical spine pathology. Presence of pain in the elbow, wrist, or hand. Clinical diagnosis of rotator cuff-related shoulder pain or frozen shoulder. Medical diagnosis of cardiovascular, rheumatologic, or neurological disorders. Pregnancy. Cognitive impairment. Concurrent physiotherapy treatment during the study period. Use of analgesic or anti-inflammatory medication within 24 hours prior to study assessments.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | From enrollment to the end of treatment at 8 weeks
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), an 11-point numerical rating scale ranging from 0 ("no pain") to 10 ("worst imaginable pain"). The NPRS has demonstrated adequate test-retest reliability, with intraclass correlation coefficients (ICC) ranging from 0.63 to 0.92, and strong internal consistency, with Cronbach's alpha values between 0.84 and 0.98, as previously reported in studies evaluating its psychometric properties (Stratford & Spadoni, 2001; Jensen & McFarland, 1993; Jensen et al., 1986)

SECONDARY OUTCOMES:
Shoulder disability | From enrollment to the end of treatment at 8 weeks
  Shoulder disability will be assessed using the Spanish version of the Shoulder Pain and Disability Index (SPADI), a self-reported questionnaire designed to measure shoulder pain and functional limitations through 13 items originally developed by Williams et al. (1995). The instrument has demonstrated the ability to discriminate between patients who improve and those who worsen (Roy et al., 2009), and its Spanish cross-cultural adaptation preserves the original structure and psychometric properties, providing a reliable and valid patient-reported outcome measure suitable for both clinical practice and research (Membrilla-Mesa et al., 2015)
External rotation strength | From enrollment to the end of treatment at 8 weeks
  Isometric external rotation strength of the shoulder will be measured using the MicroFET 2 MT Digital Handheld Dynamometer (Hoggan Health Industries, West Draper, UT). Handheld dynamometry has shown good to excellent intra-examiner reliability for isometric shoulder strength assessment, with intraclass correlation coefficients ranging from 0.87 to 0.99, according to prior studies evaluating its reproducibility in clinical and research settings (McLaine et al., 2016; Holt et al., 2016)
Hand grip strength | From enrollment to the end of treatment at 8 weeks
  Hand grip strength will be measured using a Jamar handheld dynamometer (Sammons Preston Rolyan, Bolingbrook, IL), a device widely recognized for its robustness and reproducibility. This instrument has demonstrated good to excellent intra-examiner reliability for isometric grip strength outcomes, with intraclass correlation coefficients ranging from 0.85 to 0.98 in previous validation studies (Roberts et al., 2011)
Shoulder mobility | From enrollment to the end of treatment at 8 weeks
  Shoulder range of motion will be assessed for flexion, abduction, external rotation at 0°, external rotation at 90°, and internal rotation at 90° of abduction using a validated smartphone inclinometer application (Plaincode Software Solutions, Gunzenhausen, Germany). This tool has shown excellent inter-examiner reliability and validity in symptomatic individuals, with intraclass correlation coefficients greater than 0.80 for shoulder mobility measurements (Werner et al., 2014)
Health-related quality of life | From enrollment to the end of treatment at 8 weeks
  Health-related quality of life will be measured using the Short Form-12 Health Survey (SF-12), which evaluates eight dimensions of perceived physical and mental health. This questionnaire has been widely validated across diverse populations and has consistently demonstrated strong reliability and construct validity for assessing global functional health status (Ware et al., 1996)